CLINICAL TRIAL: NCT04821232
Title: Does Yoga Done To Women With Premenstrual Syndrome Affect Inflammation Parameters?: Single Blind, Randomized Controlled Trials
Brief Title: Does Yoga Done To Women With Premenstrual Syndrome Affect Inflammation Parameters?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Aysu Yıldız Karaahmet, Principal Investigator, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: pmsyoga
Record Dates: First submitted 2021-02-11; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Sendrom; yoga; midwifery student
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: single blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The research data had blinded the statistician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): Students in the intervention group will be given a total of 120 minutes out of 40 minutes, and 24 sessions of yoga for 8 weeks, 3 days a week. The researcher who will make yoga with each student will be sent videos on the online platform, including a yoga introduction and a full yoga session with the students after a yoga session. The students were asked to do yoga 3 times a week in accordance with the video and the researcher will be called twice a week to get information about the process. Content of education;
  1. Breath Awareness Training (10 minutes)
  2. Asanas (20 minutes) I. Don't bend sideways in Mountain Pose ii. Warrior Pose iii. Bridge Pose iv. Happy Baby Pose
  v. Fixed Butterfly / Angel Pose vi. Wide sitting in Angel Pose vii. Cat Pose Tiger Breath viii. Cow-downward dog, ix. Plank x. Cobra c. Mudra and meditation (10 minutes) will be practiced.
  Interventions: Other: yoga; Other: Routin control
- Control groups (Other): No intervention will be applied to students in the control group.
  Interventions: Other: Routin control

INTERVENTIONS:
Other: yoga — Content of education;
  1. Breath Awareness Training (10 minutes)
     Students will be checked on a routine basis
  2. Asanas (20 minutes) I. Don't bend sideways in Mountain Pose ii. Warrior Pose iii. Bridge Pose iv. Happy Baby Pose
  v. Fixed Butterfly / Angel Pose vi. Wide sitting in Angel Pose vii. Cat Pose Tiger Breath viii. Cow-downward dog, ix. Plank x. Cobra c. Mudra and meditation (10 minutes) will be practiced.
  Arms: interventional
Other: Routin control — Students will be checked on a routine basis

SUMMARY:
The menstrual cycle is one of the most important signs of a functioning reproductive system in women, but sometimes this cycle is associated with signs and symptoms that cause physical and psychological problems for women.

Considering the high prevalence of PMS among women and the complications of this syndrome on work performance, social and interpersonal relationships and family, and its role in limiting education, social and economic progress in society, 8 weeks of online yoga exercises given online to female students were helpful in reducing PMS symptoms The aim was to evaluate the efficacy and effect on inflammation parameters. The study was planned as an interventional, single-blind, randomized controlled study. The sample size of this study was calculated based on the latest research available on the effect of exercise on PMS (Kamalifard et al.2017). A power analysis was performed in student PMS scores between exercise and control groups and to expect a difference of 80% strength and α = 0.50 and 30%. 80% power (1 - ß) minimum 18 students for each group, total 36 students will be included in the sample.

DETAILED DESCRIPTION:
The menstrual cycle is one of the most important signs of a functioning reproductive system in women, but sometimes this cycle is associated with signs and symptoms that cause physical and psychological problems for women.

Considering the high prevalence of PMS among women and the complications of this syndrome on work performance, social and interpersonal relationships and family, and its role in limiting education, social and economic progress in society, 8 weeks of online yoga exercises given online to female students were helpful in reducing PMS symptoms The aim was to evaluate the efficacy and effect on inflammation parameters. The study was planned as an interventional, single-blind, randomized controlled study. The sample size of this study was calculated based on the latest research available on the effect of exercise on PMS (Kamalifard et al.2017). A power analysis was performed in student PMS scores between exercise and control groups and to expect a difference of 80% strength and α = 0.50 and 30%. 80% power (1 - ß) minimum 18 students for each group, total 36 students will be included in the sample.

The researcher will provide brief information about the scope of the research by interviewing the students who meet the case selection criteria online. Verbal and written consents of the "Informed Consent Form" will be obtained (written consents will be sent to the researcher online). Female students who accepted to participate in the study were given the "Data Collection Form" (see Annex: 1), "Beck Depression Inventory" (APPENDIX: 2), Visual Pain Scale (VAS) (see APPENDIX: 3) and PMS for 3 cycles. Scale (see Annex: 4) will be applied using the online data collection method. Students who meet the sample selection criteria will be randomly allocated to the intervention and control group by the method of computer-assisted randomization (www.randomizer.org). In order to ensure blindness, randomization and random distribution of the participants to the groups will be done by a researcher and will not be shared with other researchers. and Body Mass Index will be calculated. CRP, Procalcitonin, sedimentation, Interleukin (IL) -2, IL-4, IL-6, IL-10, IL-12, and interferon from all participants on the day of the highest VAS score (the day when symptoms peak) and the day when symptoms were highest. (IFN gamma), TNF alpha and PMS scale will be taken. Students in the intervention group will be given a total of 120 minutes out of 40 minutes, and 24 sessions of yoga for 8 weeks, 3 days a week. The researcher who will make yoga with each student will be sent videos on the online platform, including a yoga presentation and a full yoga session with the students after a yoga session. The students were asked to do yoga 3 times a week in accordance with the video and the researcher will be called twice a week to get information about the process.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-35
* To be of reproductive age,
* Not giving birth before, Healthy women with regular menstrual periods (those who have bleeding between menstrual cycles for 3-8 days for 21-35 days),
* To be an undergraduate student,
* AcOG PMS criteria (according to ACOG diagnostic criteria; women with at least one premenstrual syndrome and symptoms in at least three consecutive cycles)

Exclusion Criteria:

* Having a regular yoga history for 3 months before and during the workout;
* Having a chronic disease (Endocrine, DM, Heart diseases, psychiatric illness) Oral contraceptive use
* To have a physical problem that prevents him from doing yoga asanas
* Over cyst and PICOS
* Get a score lower than 110 from the total scale score according to the PMS scale score
* Over 10 in Beck Depression Inventory, Students with a history of gynecological surgery were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premestrual sendrom
Enrollment: 36 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Standardized cross-sectional rating scales | Change from Baseline PMS scale at 2 months
  premenstrual syndrome scale
Standardized cross-sectional rating scales | Change from Baseline Beck Depression Inventory scale at 2 months
  Beck Depression Inventory
Standardized cross-sectional rating scales | Change from VAS Inventory scale at 2 months
  VISUAL ANALOG SCALE(VAS)

SECONDARY OUTCOMES:
effect on blood parameters | Change from CRP parameters at 2 months
  CRP,from all participants on the day the highest score on VAS was obtained (the day when symptoms peak) and the day when symptoms were highest
effect on blood parameters | Change from sedimentation parameters at 2 months
  sedimentation,from all participants on the day the highest score on VAS was obtained (the day when symptoms peak) and the day when symptoms were highest
effect on blood parameters | Change from progesterone parameters at 2 months
  progesterone from all participants on the day the highest score on VAS was obtained (the day when symptoms peak) and the day when symptoms were highest
effect on blood parameters | Change from estrogen parameters at 2 months
  estrogen from all participants on the day the highest score on VAS was obtained (the day when symptoms peak) and the day when symptoms were highest

CONTACTS AND LOCATIONS:
Overall Officials: Aysu Yıldız Karaahmet, Phd.Student, Principal Investigator — Halic University; Fatma Sule Tanrıverdi, PhD student, Principal Investigator — Halic University; Murat Ekmez, Dr, Study Director — Health Sciences University-Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Sultanbeyli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: until data is collected